CLINICAL TRIAL: NCT03806166
Title: Short or Long Antibiotic Regimes in Orthopaedics (SOLARIO): A Randomised Open Label Multi-Centre Clinical Trial
Brief Title: Short or Long Antibiotic Regimes in Orthopaedics
Acronym: SOLARIO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oxford University Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Matthew Scarborough, Principle Investigator, Consultant in Clinical Infection., Oxford University Hospitals NHS Trust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRAS No. 244229; PID 13859 (Other: Oxford University Hospitals NHS Foundation Trust)
Record Dates: First submitted 2019-01-11; First posted 2019-01-16 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2024-12

CONDITIONS: Osteomyelitis; Prosthetic Joint Infection; Diabetic Foot
MeSH Terms: conditions — Osteomyelitis; Diabetic Foot

STUDY DESIGN:
Intervention Model Description: Non-inferiority randomised controlled trial
Who Masked: Outcomes Assessor
Masking Description: Ascertainment of the primary outcome (treatment failure) will be undertaken by an independent committee of specialists, using redacted participant clinical records, who will remain unaware of the treatment allocation of the participant, and who will ascertain treatment failure according to established objective criteria.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Shorter Systemic Antibiotics (Experimental): Participants will receive local antibiotic therapy at the time of surgery, followed by one week or less of systemic antibiotic therapy, for bone and joint infection.
  Interventions: Other: Shorter Systemic Antibiotics
- Long Systemic Antibiotics (Active Comparator): Participants will receive local antibiotic therapy at the time of surgery, followed by four weeks or more of systemic antibiotic therapy (standard treatment recommended by international guidelines), for bone and joint infection.
  Interventions: Other: Standard treatment

INTERVENTIONS:
Other: Shorter Systemic Antibiotics — Reduced duration of post-operative systemic antibiotic therapy
  Arms: Shorter Systemic Antibiotics
Other: Standard treatment — Standard duration of systemic antibiotic treatment
  Arms: Long Systemic Antibiotics

SUMMARY:
Research question: If adults with bone or joint infection have local antibiotic therapy, can they do without prolonged treatment with antibiotics by mouth (oral) or injection?

Adults with bone or joint infections are usually given long courses of oral antibiotics or into a vein (intravenous) following surgery. It is also safe to give antibiotics directly into the bone or joint at the time of surgery: this is called local antibiotic therapy. This study investigates whether using local antibiotic therapy would allow shorter courses of oral or intravenous antibiotics, in order to limit antibiotic resistance, side effects and cost.

This study compares short against long courses of oral or intravenous antibiotics for adults who have been given appropriate local antibiotic therapy to treat bone or joint infection. Patients who can take part will be randomly divided into two groups within 7 days of surgery. One group will stop oral or intravenous antibiotics, while the other group will continue for 4 weeks or more (standard treatment).

Adults with bone and joint infections who have already had surgery and local antibiotic therapy will be invited. Patients will not take part if they need intravenous antibiotics for another reason, or if their infection is caused by bacteria resistant to the antibiotic(s) used in their local antibiotic therapy.

Main measurement: how many patients' infections return within 12 months after surgery. This will be decided by a group of doctors who do not know what treatment the patient received.

Other important measurements: serious adverse events; side-effects; quality of life; cost of treatment.

Patients will be asked questions at their usual clinic visits, and will be given a questionnaire at the start of treatment and 1 year later.

DETAILED DESCRIPTION:
Using antibiotics wisely, only when and where they are really needed, is important to prevent superbugs emerging. At the moment, bone and joint infections are usually treated by a combination of surgery and antibiotics. Traditionally, treatment relies on several weeks of antibiotics as tablets or injections (systemic antibiotics), but these can sometimes cause problems.

It is now possible to administer local antibiotics at the time of surgery directly to the site of infection. This allows much higher levels of the antibiotic to be delivered, for days or weeks, following surgery. Therefore, this study will investigate whether local antibiotics with a shorter course of systemic antibiotics can treat bone and joint infections as effectively as local antibiotics with a prolonged course of systemic antibiotics (usual treatment). If so, it may be possible to reduce antibiotic side effects, help to prevent antibiotic resistant bacteria emerging and limit overall treatment costs.

Patients who agree to participate in this study will be allocated at random to two treatment strategies after surgery for bone and joint infection.

One group of patients will be treated with local antibiotics and a long course of systemic antibiotics, which is the usual treatment: this is the 'long group'.

The other group will be treated with local antibiotics and a short course of systemic antibiotics: this is the 'short group' whose treatment differs from the current usual treatment.

Patients will be involved in the study for one year, and infection recurrence will be assessed at the time of routine clinic review up to 12 months after surgery. Whether or not treatment has been successful will be assessed by an independent committee of specialists, who will remain unaware of the patient's allocated treatment strategy.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent
2. Aged 18 years or over
3. Presenting with an orthopaedic infection, defined by one or more of the following criteria:

   1. localised pain, OR
   2. localised erythema, OR
   3. temperature ≥ 38.0 C, OR
   4. a discharging sinus or wound
4. Undergoing surgical treatment for the infection
5. Locally administered antibiotic(s) at the site of orthopaedic infection
6. Has received <= 7 days of systemic antimicrobial therapy after surgery
7. Would ordinarily be managed with a prolonged course (>= 4 weeks) of systemic antibiotic(s)
8. Specimens for microbiological analysis taken at index surgery

Exclusion Criteria:

Surgical exclusion criteria

1. The index operation was not a definitive procedure with the aim of eradicating infection:

   1. Primary closure has not been achieved, or
   2. Re-look surgery is planned
2. The index operation involved implant retention (e.g. DAIR)

   Microbiological exclusion criteria
3. Any identified micro-organisms from operative specimens from the site of incident infection are fully resistant to the local antibiotic(s) administered at the site of infection

   Medical exclusion criteria
4. Other infection necessitating additional systemic antibiotic treatment beyond 7 days after surgery, such as Staphylococcus aureus bacteraemia, psoas abscess, discitis or bacterial endocarditis
5. If the patient is in a clinical trial involving an Investigational Medicinal Product (IMP) related to infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2019-02-21 (Actual); Primary Completion 2024-12-04 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Definitive treatment failure (infection recurrence) | 12 months from the time of surgery for bone or joint infection
  Proportion of participants in each treatment group experiencing definitive treatment failure (infection recurrence), ascertained by an independent committee of experts unaware of the treatment allocation of the participant, according to established criteria.

SECONDARY OUTCOMES:
Possible or probable treatment failure | 12 months from the time of surgery for bone or joint infection
  Proportion of participants in each treatment group experiencing clinical features suggesting possible or probable infection recurrence, not meeting the definition for definitive treatment failure, determined by an independent committee of experts unaware of treatment allocation, where microbiological culture is not done or is negative. Ascertainment is based on established clinical criteria associated with, but not diagnostic of, orthopaedic infection.
Serious Adverse Events | 12 months from the time of surgery for bone or joint infection
  Proportion of participants in each treatment group experiencing Serious Adverse Events including mortality
Antibiotic side effects | This will be assessed at baseline (pre-randomisation, at <7 days of treatment), 6 weeks and 3 months from the time of surgery for bone or joint infection
  Proportion of participants in each treatment group experiencing possible side-effects from systemic antibiotic treatment, adjusted for severity on a 3-point scale
Quality of life measured by EuroQol 5 Dimensions 5 Levels Score and EuroQol Visual Analogue Score | At baseline and 12 months from the time of surgery for bone or joint infection
  EQ-5D-5L score distribution across 5 dimensions (mobility, self-care, ability to complete usual activities, pain or discomfort, anxiety or depression) for participants, ranging from 1 (worst) to 5 (best) for each dimension. EQ-VAS score distribution for participants, for self-reported health state, ranging from 0 (worst) to 100 (best).

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Scarborough, Principal Investigator — Oxford University Hospitals
Locations (23):
- Universitaetsklinikum Regensburg, Regensburg, Germany
- Hospital San Antonio, Porto, Portugal
- Parc de Salut Mar, Barcelona, Spain
- United Kingdom (20):
  - University Hospitals Dorset, Poole, Dorset
  - Southampton General Hospital, Southampton, Hampshire
  - Wrightington Hospital, Wigan, Lancashire
  - Barts and the Royal London Hospitals, London, London
  - Royal National Orthopaedic Hospital, Stanmore, London
  - The Robert Jones & Agnes Hunt Hospital, Gobowen, Oswestry
  - Bone Infection Unit, Nuffield Orthopaedic Centre, Oxford, Oxfordshire
  - Great Western Hospital, Swindon, Wiltshire
  - University Hospitals Birmingham, Birmingham
  - Blackpool Teaching Hospitals NHS Foundation Trust, Blackpool
  - Brighton & Sussex University Hospitals NHS Trust, Brighton
  - Royal Liverpool Hospitals, Liverpool
  - London North West Healthcare NHS Trust, London
  - Imperial College Healthcare NHS Trust, London
  - Manchester University NHS Foundation Trust, Manchester
  - Northumbria Healthcare NHS Foundation Trust, Newcastle
  - Nottingham University Hospitals NHS Trust, Nottingham
  - The Rotherham NHS Foundation Trust, Rotherham
  - Salisbury NHS Foundation Trust, Salisbury
  - The Mid Yorkshire Hospitals NHS Trust, Wakefield

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dudareva M, Kumin M, Vach W, Kaier K, Ferguson J, McNally M, Scarborough M. Short or Long Antibiotic Regimes in Orthopaedics (SOLARIO): a randomised controlled open-label non-inferiority trial of duration of systemic antibiotics in adults with orthopaedic infection treated operatively with local antibiotic therapy. Trials. 2019 Dec 9;20(1):693. doi: 10.1186/s13063-019-3832-3. PMID 31815653